CLINICAL TRIAL: NCT06852820
Title: A Pilot Study of 68Ga-PSMA-11 PET-directed Radioligand Therapy in Patients With Metastatic Hepatocellular Carcinoma (HCC)
Brief Title: 68Ga-PSMA-11 PET-directed Radioligand Therapy in Metastatic Hepatocellular Carcinoma (HCC)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Melissa Lumish (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Melissa Lumish, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE7224
Record Dates: First submitted 2025-02-25; First posted 2025-02-28 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Liver Cancer; Hepatocellular Carcinoma; Metastatic Liver Cancer
Keywords: Ga-PSMA-11
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Pluvicto

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lu-PSMA-617 (Experimental): Participants will receive 177Lu-PSMA-617 7.4 GBq (200 mCi) once every 6 weeks. 177Lu-PSMA-617 is a radiopharmaceutical which will be administered intravenously (IV).
  Interventions: Drug: Lu-PSMA-617

INTERVENTIONS:
Drug: Lu-PSMA-617 — Given IV

SUMMARY:
The purpose of this study is to look at the effects (good and bad) of a drug called 177Lu-PSMA-617 (also known as the study drug) when given to participants who have prostate specific membrane antigen (PSMA) positive liver cancer.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the third leading cause of cancer-related deaths worldwide, with more than 900,000 newly diagnosed cases and approximately 830,000 deaths in 2020. Surgical resection and liver transplantation are potential curative options for patients with early-stage HCC. However, most patients present with metastatic and/or unresectable disease and systemic treatment is the only therapeutic option for these patients.

Although several ICI-based combination therapies have recently extended survival for many patients with HCC, biomarker-directed strategies are limited for this disease. Prostate Specific Membrane Antigen (PSMA) is a protein that is expressed in prostate cells and overexpressed in prostate cancer and is accepted as a valuable theragnostic (combined diagnostic and therapeutic) target in metastatic castration-resistant prostate cancer. 68Ga-PSMA-11 PET (PSMA PET) is now utilized to select patients with metastatic prostate cancer for PSMA-directed therapy with 177Lu-PSMA-617. PSMA is now known to be expressed in a variety of solid tumors, including HCC, specifically in the neovasculature associated with solid tumors. However, there is a lack of data exploring whether there is a role for PSMA-directed therapy in non-prostate solid tumors.

Investigator performed PSMA IHC on 148 HCCs from surgical resection or liver explant specimens from patients at the Mayo Clinic, and 90% of HCCs showed PSMA immunostaining localized to the tumor endothelium. More than 50% of HCCs showed 31-100% PSMA immunostaining by area. In several cases, the normal liver background did show faint canalicular staining, highlighting the need to distinguish between normal tissue and tumor-associated expression.

In a similar study using immunohistochemistry (IHC) to evaluate PSMA expression in HCC, 79.2% of tumors showed high levels of PSMA expression at any location, with the majority of this expression occurring in a neovascular staining pattern (89.9%). One patient underwent imaging with PSMA PET which demonstrated intense and heterogeneous PSMA uptake in the HCC tumor.

Several additional reports have demonstrated that PSMA expression in HCC can be detected noninvasively by PSMA PET.20,21 Our group at Mayo Clinic prospectively evaluated PSMA uptake using Ga-PSMA PET in patients with treatment-naïve HCC. In 31 patients, 39 lesions were identified. In this study, 64% had high PSMA uptake (grade 3 or 4) and 36% had low PSMA uptake (grade 1 or 2). It is expected that PSMA uptake will be much higher in patients with advanced HCC. PSMA PET has been compared with MRI for detection of HCC and had similar efficacy to MRI in a cohort of 19 patients. Similarly, a meta-analysis of 6 studies including 126 patients imaged with PET/CT or PET/MRI with PSMA-targeting radiopharmaceuticals in patients with newly diagnosed or recurrent HCC showed a detection rate of greater than 85%.These studies clearly suggest that targeting PSMA could be an attractive target in patients with advanced HCC.

The VISION study was a phase 3 trial investigating the efficacy and safety of 177Lu-PSMA-617 (Lu-177 vipivotide tetraxetan) with standard of care in patients with previously treated metastatic castration-resistant prostate cancer who were identified as PSMA PET-positive. Similarly, the phase III PSMAfore study of Lu-177 vipivotide tetraxetan demonstrated improvement in radiographic progression-free survival in patients with metastatic castration-resistant prostate cancer after prior treatment.

In HCC, a recent preclinical study demonstrated that radioligand therapy using [177Lu]Lu-PSMA-617 and [177Lu]Lu-EB-PSMA-617 effectively suppressed tumor growth and prolonged survival time in PSMA-positive HCC xenograft mice. However, this strategy has not been prospectively utilized in patients with HCC after first-line therapy. There is limited clinical data examining the role of PSMA radioligand therapy in HCC. One study included 2 patients with no other systemic therapy options available and demonstrated insufficient tumor radiation dosing by intratherapeutic SPECT/CT-based dosimetry after only a single cycle of therapy. This data is limited by the short treatment course of only 1 cycle, which was inadequate to induce a response, small sample size, and heavy pre-treatment.

Although the pattern of PSMA expression in HCC is distinct from that in prostate cancer, there is evidence from tyrosine kinase inhibitor (TKI) efficacy that targeting the neovasculature via inhibition of angiogenesis in the local tumor environment can limit tumor growth and improve survival.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically, cytologically or radiographically confirmed hepatocellular carcinoma by LI-RADS30 with metastatic and/or unresectable disease.
* Participants must have received one prior line of systemic therapy for the treatment of metastatic and/or unresectable HCC including anti-PD-L1 therapy. Participants will be enrolled at the time of progression on first-line therapy for metastatic and/or unresectable disease.
* Age >18 years. Because no dosing or adverse event data are currently available on the use of 177Lu-PSMA-617 (Lu-177 vipivotide tetraxetan) in participants <18 years of age, children are excluded from this study.
* ECOG performance status 0 or 1.
* Participants must have normal organ and marrow function as defined below:

Absolute Neutrophil Count ≥ 1,500/mcL. Hemoglobin > 9 g/dL. Platelet count ≥ 75,000/mcL. Serum creatinine ≤ 1.5 x institutional upper limit of normal or CrCl ≥60 mL/min using the Cockroft-Gault formula for participants with creatinine levels >1.5 ULN.

Child-Pugh class A or B7.

* At least one target lesion measurable by RECIST 1.1 criteria.
* PSMA-PET demonstrating PSMA PET positive lesion (higher uptake in the tumor compared with background liver uptake).
* Participants must have the ability to understand and the willingness to sign a written informed consent document.
* Participants of childbearing age are using an appropriate method of contraception.

Exclusion Criteria:

* Participants receiving any other investigational agents.
* Subject has received investigational therapy within 4 weeks or within 5 half-lives of the therapeutic agent (whichever is shorter).
* Ongoing grade 3 or higher toxicity from prior anticancer systemic therapy.
* Prior treatment with Y90 radioembolization for hepatocellular carcinoma.
* Participants who have undergone major surgery within 3 months of screening and have not adequately recovered.
* Known additional malignancy that currently requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Participants with untreated brain metastases and/or carcinomatous meningitis will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Participants with previously treated brain metastases may participate provided they are stable without evidence of new or enlarging brain metastases and are not using steroids for at least 7 days prior to trial treatment.
* Participants with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Participants with known psychiatric or substance use disorders that would interfere with cooperation with the requirements of the trial, in the opinion of the treating investigator.
* Subject is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 7 months for females and 14 weeks for males after the last dose of trial treatment. Pregnant or breastfeeding women are excluded from this study because 177Lu-PSMA-617 has not been previously studied in this population and the potential for teratogenic or abortifacient effects are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to the treatment of the mother with 177Lu-PSMA-617, breastfeeding should be discontinued if the mother is treated with 177Lu-PSMA-617. These potential risks may also apply to 68Ga-PSMA-11 used in this study.
* Subject has received live vaccine within 30 days prior to the first dose of trial treatment.
* Subject with recent variceal bleeding, gastrointestinal bleeding or high risk of bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with PSMA-Avid Lesions on PET Imaging (≥50%) | 12 weeks post intervention
  Study is feasible if at least 1 PSMA-PET positive lesion is identified in at least 50% of the participants in this cohort
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 240 days post treatment

SECONDARY OUTCOMES:
Progression free survival (PFS) | 24 weeks post intervention
  PFS will be estimated using Kaplan-Meier method
Median overall survival(OS) | 52 weeks post intervention
  OS will be estimated using Kaplan-Meier method
Objective response rate(ORR) | 12 weeks post intervention
  The ORR will be estimated based on the number of participants with clinical response using a binomial distribution and its confidence interval will be estimated using Wilson's method
Clinical benefit rate | 12 weeks post intervention
  Clinical benefit rate as defined as proportion of participants with objective responses or stable disease at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Lumish, MD, Principal Investigator — Case Comprehensive Cancer Center, University Hospitals Cleveland Medical Center
Locations (1):
- Case Comprehensive Cancer Center, University Hospitals Cleveland Medical Center, Seidman Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
This is an investigator initiated trial and University hospital will have the access to individual level data